CLINICAL TRIAL: NCT06222255
Title: The Safety and Efficacy of Transanal Irrigation in Patients With Sleep Disturbance From Low Anterior Resection Syndrome After Rectal Cancer Surgery: A Multicenter Prospective Randomized Controlled Trial (TraLARS)
Brief Title: The Safety and Efficacy of Transanal Irrigation in Patients With Sleep Disturbance From Low Anterior Resection Syndrome After Rectal Cancer Surgery (TraLARS)
Acronym: TraLARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2310-121-1479
Record Dates: First submitted 2024-01-08; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer; Insomnia; Sleep Disorder
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loperamide group (No Intervention): The group only takes loperamide in the evening.
- Loperamide + Transanal irirgation group (Experimental): The group takes Loperamide in the evening and undergoes Transanal irrigation before bedtime.
  Interventions: Procedure: Transanal Irrigation (TAI)

INTERVENTIONS:
Procedure: Transanal Irrigation (TAI) — The combination of transanal irrigation (TAI) and Loperamide (Lopmin®) involves administering Loperamide orally, with a daily dosage of 2 mg for males (2 tablets once daily) and 1 tablet for females (1 tablet once daily). This is complemented by the use of TAI, a method in which patients self-administer water into the rectum through an enema, aiming to enhance bowel management and potentially alleviate symptoms associated with LARS (Low Anterior Resection Syndrome).
  Arms: Loperamide + Transanal irirgation group

SUMMARY:
The preservation surgery of the anal sphincter muscle has become the standard procedure in the treatment of rectal cancer and, thanks to advancements in surgical techniques, can now be performed for tumors located closer to the anus. This method allows patients to avoid a permanent artificial anus, maintaining continuity of the intestines and enabling bowel movements through the anus, making it a highly preferred procedure. Furthermore, advancements in various tumor treatments have led to improved long-term survival rates.

Preservation surgery of the anal sphincter muscle is commonly used in the treatment of rectal cancer, resulting in approximately 90% of patients experiencing changes in bowel habits after surgery. These changes include characteristic diarrhea, urgent bowel movements, frequent bowel movements, and fecal incontinence, collectively known as Anterior Resection Syndrome (ARS). Particularly in the case of low rectal cancer, it often manifests as Low Anterior Resection Syndrome (LARS). These symptoms are most severe immediately after surgery, generally persisting in a significant degree for 1-2 years, with some improvement over time. However, for many patients, LARS remains a lifelong challenge, significantly impacting their quality of life. Nighttime symptoms of LARS, in particular, have a profound effect on sleep quality, potentially leading to a decline in overall quality of life.

Currently, there is no definitive method to completely cure LARS, and the available approaches focus on empirical treatments or short-term symptom control using medications such as loperamide.

Loperamide directly affects the neuromuscular system of the intestine, reducing its motility. This prolongs the time food stays in the intestine, allowing sufficient absorption of moisture and electrolytes, consequently reducing symptoms of diarrhea. Loperamide is available in two forms: loperamide oxide and loperamide hydrochloride. While loperamide oxide products like Arestal® were prescribed by doctors until August 2017, the approval was revoked, leaving loperamide hydrochloride as the only form used domestically. It comes in a single product containing 2 mg of loperamide hydrochloride and a combination product with 0.25 mg of loperamide hydrochloride, a sterilizing agent in the intestine (e.g., acrylonitrile, berberine), and an antispasmodic.

Transanal irrigation (TAI) is a method where patients self-administer water into the rectum through an enema, physically cleansing the anus and rectum. This technique is often used for patients with chronic constipation or fecal incontinence. TAI has proven beneficial, particularly in improving symptoms for patients experiencing bowel dysfunction following sphincter-preserving surgery, especially for those who underwent low anterior resection.

However, there is currently no research on the utility and safety of TAI for LARS patients, specifically addressing whether it can improve the nighttime symptoms associated with LARS syndrome and enhance sleep quality. Therefore, this study aims to investigate the impact of TAI on the quality of sleep in patients with nighttime symptoms of LARS syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years and above.
2. Patients who have undergone low or ultra-low anterior resection surgery for rectal cancer (within 15cm from the anal verge).
3. Patients at least 24 months post-surgery (excluding those with incontinence, patients who have undergone postoperative cancer treatment should have completed treatment, and patients who have undergone bowel restoration surgery should be at least 6 months post-surgery, or for patients who received long-course preoperative radiotherapy, at least 18 months post-surgery).
4. Patients evaluated with a major LARS score who also have an ISI score of 3 or 4.
5. Patients who comprehend and have the ability to participate in this clinical trial.

Exclusion Criteria:

1. Patients currently taking medication for LARS within the last month.
2. Patients with a history of prior surgery for colorectal cancer.
3. Patients with recurrent colorectal cancer.
4. Patients with concomitant metastatic colorectal cancer.
5. Patients requiring permanent colostomy.
6. Patients who have undergone postoperative cancer radiation therapy.
7. Patients with underlying conditions not controlled by internal medical treatment.
8. Patients with inflammatory bowel disease (IBD).
9. Patients with symptoms of constipation or diarrhea not controlled by medication.
10. Patients with preoperative symptoms of fecal incontinence.
11. Patients allergic to the investigational drug.
12. Patients deemed unsuitable for clinical trial participation by the principal investigator and study personnel.
13. Patients with ISI scores of 1 or 2.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The LARS (Low Anterior Resection Syndrome) Score with Night symptoms | 4 weaks
  A survey was conducted, scoring patients' symptoms related to LARS.

SECONDARY OUTCOMES:
Insomnia Severity Index score in Korean Validation | 4 weaks
  A survey was conducted, scoring patients' symptoms related to Insomnia
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - C30 | 4 weaks
  A survey was conducted, scoring patients' symptoms related to LARS and Quality of Life
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - CR29 | 4 weaks
  A survey was conducted, scoring patients' symptoms related to LARS and Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongro-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided